CLINICAL TRIAL: NCT01710865
Title: Evidence Based Effectiveness of Pit and Fissure Sealants Applied By Students and Paediatric Dentists After (Three) Five Years.
Brief Title: Effectiveness of Two Sealant Materials Over 5 Years
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 041386
Record Dates: First submitted 2012-07-24; First posted 2012-10-19 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Caries
Keywords: Caries prevention; pit and fissure sealants
MeSH Terms: conditions — Van der Woude syndrome | interventions — Ultra Seal XT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultraseal Sealant (Experimental): Both Ultraseal XT Hydro and Ultraseal XT Plus will be applied on patients.
  Interventions: Other: Ultraseal Sealant

INTERVENTIONS:
Other: Ultraseal Sealant — This is a newly developed hydrophilic sealant material.
  Other Names: Ultraseal XT Hydro
Other: Ultraseal Sealant — This is a previously existing hydrophobic sealant material.
  Other Names: Ultraseal XT Plus

SUMMARY:
The purpose of this study is to assess the effectiveness of a new hydrophilic sealant (Ultraseal XT Hydro) compared to the previously existing hydrophobic sealant materials (Ultraseal XT Plus) which requires prime and dry to dry the tooth surface.

DETAILED DESCRIPTION:
The new hydrophobic sealant material eliminates the step of prime and drying the tooth which prevents from over drying the tooth surface and decreases chair time, which is important when working with children. The null hypothesis is that there is no difference between the materials. The alternate hypothesis is that the Ultraseal XT Hydro is a better material.

ELIGIBILITY:
Inclusion Criteria:

* Children that are at a high risk of developing caries.

Exclusion Criteria:

* Children that already have sealants or do not need them.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Changes in retention of sealants from baseline to five years | Baseline and every year (baseline to five years)
  The assessment of the retention of sealants (intact, partially lost, completely lost) will be carried out every year for 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sahza Hatibov-Kofman, D.D.S.FRCD, Principal Investigator — Division of Orthodontics and Paediatric Dentistry
Locations (1):
- Children's Clinic at Western University, London, Ontario, Canada